CLINICAL TRIAL: NCT04538482
Title: Determining the structural-and Functional-level Effects of Diet-specific Interventions on the Gut-microbiota of a Diverse Sample of Southern United States Adults
Brief Title: DASH INtervention to INvestigate the Gut
Acronym: DINING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MCC-21224; R01CA253219 (NIH)
Record Dates: First submitted 2020-08-29; First posted 2020-09-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Microbiota; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DASH Diet (Experimental): calorie-restricted DASH diet (25% fat; 57% carbohydrate; 18% protein; 34 g fiber)
  Interventions: Behavioral: DASH Diet
- standard American diet (Active Comparator): calorie-restricted standard American diet (35% fat; 51% carbohydrate; %15 protein; 14 g fiber)
  Interventions: Behavioral: standard American diet

INTERVENTIONS:
Behavioral: DASH Diet — Participant will receive foods following the DASH dietary pattern for 28 days.
  Arms: DASH Diet
Behavioral: standard American diet — Participants will receive foods following the standard American diet for 28 days.
  Arms: standard American diet

SUMMARY:
The study investigators will recruit a generally healthy sample of 112 black and white adults from Birmingham, AL to participate in a 28-day randomized, controlled feeding study. Participants will be randomized to receive either the DASH diet or a standard American diet. All meals will be provided by the study. Fecal samples will be collected at multiple time points before, during, and after the dietary intervention and will be analyzed using PCR to amplify the V4 region of the 16S rRNA gene and to sequence bases using the MiSeq platform. Sequenced data will then be analyzed using QIIME. The investigators hypothesize that participants receiving the DASH diet will have a greater increase in alpha diversity and greater changes in abundances of CRC-associated microbes than participants receiving the standard American diet. The investigators will also evaluate functional-level markers including bile acid and short chain fatty acid (SCFA) production and inflammatory markers. If the investigator's hypothesis is supported, they expect to see reduced production of secondary bile acids (e.g., deoxycholic acid), greater SCFA production (e.g, butyrate), and reduction in gut and systemic inflammation (e.g, calprotectin, IL-6) among participants receiving the DASH diet compared to the standard American diet. The investigator's findings will provide preliminary evidence for the DASH diet as an approach for cultivating a healthier gut microbiota across racially diverse populations. These findings can impact clinical, translational, and population-level approaches for modification of the gut microbiota to reduce risk of chronic diseases like CRC.

ELIGIBILITY:
Inclusion Criteria:

* black or white race
* non-Hispanic ethnicity
* age 19-65 years
* able to travel to the UAB Bionutrition Unit daily to retrieve meals

Exclusion Criteria:

* gastrointestinal (GI) conditions i.e., irritable bowel, diverticulitis, peptic ulcers, Crohn's, GI cancers, and adenatomous polyps
* antibiotic or probiotic use in the previous 90 days
* smoking/tobacco use
* heavy alcohol consumption
* major medical conditions (e.g., renal disease, diabetes, cancer

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in alpha diversity | baseline - day 28
  The investigators will assess the difference in alpha diversity determined by analyzing fecal samples.
Mean change in alpha diversity | day 28 - day 42
  The investigators will assess the difference in alpha diversity determined by analyzing fecal samples.
Diet specific changes in secondary bile acids | baseline - day 28
  The investigators will calculate changes in cholic acid in milligrams
Diet specific changes in secondary bile acids | day 28 - day 42
  The investigators will calculate changes in cholic acid in milligrams
Diet-specific changes in inflammatory marker | baseline - day 28
  The investigators will calculate changes in interleukin-6 in pg/L
Diet-specific changes in inflammatory marker | day 28 - day 42
  The investigators will calculate changes in interleukin-6 in pg/L

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany L Carson, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carson TL, Buro AW, Miller D, Pena A, Ard JD, Lampe JW, Yi N, Lefkowitz E, William VP, Morrow C, Wilson L, Barnes S, Demark-Wahnefried W. Rationale and study protocol for a randomized controlled feeding study to determine the structural- and functional-level effects of diet-specific interventions on the gut microbiota of non-Hispanic black and white adults. Contemp Clin Trials. 2022 Dec;123:106968. doi: 10.1016/j.cct.2022.106968. Epub 2022 Oct 18. PMID 36265810